CLINICAL TRIAL: NCT05907057
Title: A Single Arm, Open-label Phase 3b Study to Describe the Safety and Tolerability of Ivosidenib in Combination With Azacitidine in Adult Patients Newly Diagnosed With IDH1m Acute Myeloid Leukemia (AML) Ineligible for Intensive Induction Chemotherapy
Brief Title: An Open-label Phase 3b Study of Ivosidenib in Combination With Azacitidine in Adult Patients Newly Diagnosed With IDH1m Acute Myeloid Leukemia (AML) Ineligible for Intensive Induction Chemotherapy.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Servier Affaires Médicales (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIM-95031-006; 2022-501709-11 (EudraCT Number)
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: IDH1 Mutation AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — ivosidenib; Tablets; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open-Label Ivosidenib in combination with Azacitidine (Experimental): All participants will receive both Ivosidenib and Azacitidine for a maximum of 28 cycles. Each cycle will be 4 weeks or 28 days long. Ivosidenib will be taken continuously throughout each cycle and Azacitidine will be taken only for 7 days at the beginning of each cycle.
  Interventions: Drug: Ivosidenib 500mg Oral Tablet; Drug: Azacitidine

INTERVENTIONS:
Drug: Ivosidenib 500mg Oral Tablet — Provided as tablets, taken orally as two 250mg tablets once daily.
Drug: Azacitidine — Administered subcutaneously (SC) or intravenously (IV) at a dose of 75mg/m2/day for 7 days, either consecutively on Days 1-7 or discontinuously for Days 1-5 and 8-9 of each cycle. The 7 days of administration will occur at the beginning of every 4 week-long cycle.

SUMMARY:
The purpose of this study is to learn more about the safety and efficacy of ivosidenib taken with azacitidine to treat adult patients with acute myeloid leukemia (AML) who are presenting a gene mutation called IDH1 (isocitrate dehydrogenase1 mutation-positive [IDH1m]) and cannot receive treatment with intensive chemotherapy (IC).

DETAILED DESCRIPTION:
Participants who are eligible and enroll in the study will attend a study visit on the first day of each 28-day cycle. Study visits will consist of a physical exam, blood work, electrocardiogram (ECG) and other assessments. After treatment discontinuation participants will be contacted every 12 weeks through the end of the study (currently planned for 2026) to assess survival. The study drug, Ivosidenib, will be taken once daily throughout the duration of participation in the study, and Azacitidine will only be administered for 7 days at the beginning of each 28 day cycle. If at any point ivosidenib is made available as a medical prescription at the patient's site, the patient will switch to commercial product and will continue to be followed according to the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Has untreated Acute Myeloid Leukemia (AML)
* Have a documented IDH1 R132 gene-mutated disease
* Have at least one of the following making yourself ineligible for intensive chemotherapy (IC): 75 years or older, Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 2, or any comorbidity that the investigator judges to be incompatible with IC including but not limited to severe cardiac or pulmonary disorder, creatinine clearance less than 45 mL/minute, or bilirubin greater than 1.5 times the upper limit of normal
* Has adequate hepatic (liver) and renal (kidney) function
* Female participants of reproductive potential must have a negative blood pregnancy test and must use effective contraception during treatment and for at least 6 months following treatment
* Fertile male participants with female partners of reproductive potential must use effective contraception during treatment and for at least 3 months following treatment

Exclusion Criteria:

* Has received any prior treatment for AML, with the exception of hydroxyurea or leukapheresis for white blood cell count control
* Has received prior treatment with an IDH1 inhibitor
* Is a woman who is pregnant or breastfeeding
* Has an active, uncontrolled, systemic fungal, bacterial, or viral infection (including human immunodeficiency virus [HIV], active hepatitis B (HBV), or hepatitis C virus [HCV]) without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment
* Has had significant active cardiac disease within 6 months prior to the start of study treatment, including Class III or IV congestive heart failure, myocardial infarction (heart attack), unstable angina (chest pain), and/or stroke
* Has dysphagia (difficulty swallowing), short-gut syndrome, gastroparesis (stomach paralysis), or any other condition that limits the ingestion or gastrointestinal absorption of orally administered drugs
* Has uncontrolled hypertension (high blood pressure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs) | up to week 116
  Adverse events (AEs) will be graded according to the CTCAE v5.0
Number of Serious Adverse Events (SAEs) | up to week 116
  Adverse events (AEs) will be graded according to the CTCAE v5.0
Differentiation Syndrome of Grade 2 or higher | up to week 116
Number of Adverse Events (AEs) leading to ivosidenib + azacitidine discontinuation | up to week 112
Number of Adverse Events (AEs) leading to ivosidenib + azacitidine interruption | up to week 112
Number of Adverse Events (AEs) leading to ivosidenib + azacitidine dose reduction | up to week 112
Number of Adverse Events (AEs) leading to death | up to week 116
Number of clinical laboratory anomalies assessed as Adverse Events (AEs) | up to week 116
Number of patients requiring transfusion (platelet and RBC) and the average number of units transfused | up to week 116
Rate of infections | up to week 116
  Infection rates will be summarized by classification and will include a count and proportion.
QT Prolongation event assessed as Grade 3 or higher | up to week 116

SECONDARY OUTCOMES:
Event-free survival (EFS) | up to week 116
Proportion of patients who achieve a complete remission (CR) | up to week 116
Proportion of patients who achieve complete remission plus complete remission with partial hematologic recovery rate (CR + CRh) | up to week 116
Proportion of patients who achieve complete remission plus complete remission with incomplete hematologic recovery rate (CR + CRi) | up to week 116
Duration of response (DOR) | up to week 116
Time to response (TTR) | up to week 116
Overall survival (OS) | until study closure
Quality of life (QoL), as measured by Hematologic Malignancy-Patient-Reported Outcome (HM-PRO) | up to week 116
  For patients with a baseline assessment and at least 1 post-baseline assessment that generates a score
Quality of life (QoL), as measured by Family Reported Outcome Measure (FROM-16), for caregivers and/or family | up to week 116
  For patients with a baseline assessment and at least 1 post-baseline assessment that generates a score
Health economic measures, as assessed by the 5-level EuroQol 5-Dimensions (EQ-5D-5L) | up to week 116
  For patients with a baseline assessment and at least 1 post-baseline assessment that generate a score
Average proportion of days at home | up to week 116
  Defined by subtracting the number of care days (days hospitalized or seen in an ED / oncology clinic / infusion center) from the total days of follow-up, divided by total days of follow-up

CONTACTS AND LOCATIONS:
Locations (15):
- Austria (2):
  - AKH - Medizinische Universität Wien, Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels
- France (5):
  - Institut Paoli Calmettes, Marseille, Bouches-du-Rhône
  - CHU CAEN - Hôpital de la Côte de Nacre, Caen, Calvados
  - CHU de Toulouse pt, Toulouse, Haute Garonne
  - CHU Rennes - Hopital Pontchaillou, Rennes, Ille et Vilaine
  - CHU Angers - Hôpital Hôtel Dieu, Angers, Liore
- Italy (4):
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Brescia, Brescia
  - IRCCS Istituto Scientifico Romagnolo Per Lo Studio Dei Tumori "Dino Amadori" - IRST, Meldola, Forli-Cesena
  - IRCCS Ospedale Policlinico San Martino, Genova, Genova
  - Azienda Ospedaliera di Perugia Ospedale S. Maria della Misericordia, Perugia, Perugia
- Netherlands (4):
  - Meander Medisch Centrum, Amersfoort
  - Amsterdam UMC, Amsterdam
  - Rijnstate, Arnhem
  - Universitair Medisch Centrum Groningen, Groningen

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorization in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com/

REFERENCES:
- [Derived] Vyas P, Salek S, Vives S, Recher C, Dohner H, Venditti A, Derrien H, Chatin S, De La Bigne AM, Pelouchova J, Hills R, Nier S. ALIDHE phase 3b study design: ivosidenib + azacitidine in adults with newly diagnosed IDH1 mutant acute myeloid leukemia. Future Oncol. 2025 Dec;21(29):3721-3729. doi: 10.1080/14796694.2025.2567838. Epub 2025 Nov 15. PMID 41241779